CLINICAL TRIAL: NCT06507423
Title: Study to Evaluate the Performance of the SeptiCyte LAB Test for Antibiotic Stewardship in Mesenteric Ischemia
Brief Title: Performance of the SeptiCyte LAB Test for Antibiotic Stewardship in Mesenteric Ischemia
Acronym: SPASM
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: NOVY_2024_PI_090
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Acute Mesenteric Ischemia; Sepsis Bacterial; Intra-abdominal Infection; Digestive Inflammation
Keywords: acute mesenteric schema; sepsis; septicyte; antimicrobial stewardship; intra-abdominal infection; aortic vascular surgery; surgical aortic clamping
MeSH Terms: conditions — Intraabdominal Infections; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Control group: The control group will consist of adult patients undergoing open vascular surgery for the treatment of an aortic aneurysm. This procedure requires surgical aortic clamping of variable duration, which may lead to potential ischemic events in the digestive system
  Interventions: Device: Septicyte Lab Test pre operative; Device: Septicyte Lab Test post operative
- Case: The "case" group consist of adult patients suffering from acute mesenteric ischemia who required urgent surgery
  Interventions: Device: Septicyte Lab Test pre operative; Device: Septicyte Lab Test post operative

INTERVENTIONS:
Device: Septicyte Lab Test pre operative — SeptiCyte® technology uses proprietary biomarker signatures to assess the response of a patient's immune system to infections. It provides a score which can be used to differentiate sepsis from systemic inflammatory response.
  Each included patient will received the Septicyte LAB test before and after surgery for acute mesenteric ischemia suspicion. The results will be compared to standard of care, retrospectively.
Device: Septicyte Lab Test post operative — SeptiCyte® technology uses proprietary biomarker signatures to assess the response of a patient's immune system to infections. It provides a score which can be used to differentiate sepsis from systemic inflammatory response.
  Each included patient will received the Septicyte LAB test before and after surgery for acute mesenteric ischemia suspicion. The results will be compared to standard of care, retrospectively.

SUMMARY:
This study will help determine whether the SeptiCyte LAB test can accurately differentiate between SIRS and actual infections in postoperative patients, potentially reducing unnecessary antibiotic use and improving patient outcomes in cases of acute mesenteric ischemia

DETAILED DESCRIPTION:
Introduction Early diagnosis of bacterial infections is crucial in intensive care, as conditions such as sepsis and septic shock are emergencies with high mortality rates. Conversely, Systemic Inflammatory Response Syndrome (SIRS) is a deregulated response to an insult without an infectious origin. SIRS is common post-major surgery and complicates the diagnosis between a simple inflammatory response and an actual infection. Although antibiotic therapy is undisputed in septic shock, the rise of antibiotic resistance and the lack of new antibiotics demand a judicious and well-argued prescription in probable sepsis cases. Rapid diagnostics are essential to identify patients who will benefit from empirical antibiotic therapy.

Current Diagnostic Challenges Microbiological documentation remains the gold standard for confirming sepsis or septic shock. However, the delay in obtaining standard bacteriology results poses a risk to patient survival. Biomarkers like CRP and PCT have been proposed for sepsis diagnosis, but their reliability is limited by numerous confounding factors, making them less specific.

The SeptiCyte LAB Test Recent advances in sequencing technology have made molecular biology techniques more accessible and rapid. SeptiCyte LAB is a molecular test based on the quantitative sequencing of mRNA from four genes (CEACAM4, LAMP1, PLA2G7, and PLAC8) involved in bacterial infection signaling. Studies have shown a specificity of 94% and a negative predictive value of 98.8% in ICU patients suspected of sepsis, with a threshold value above 4. These results have also been confirmed in elective esophageal surgery populations, demonstrating encouraging statistical performance.

Relevance to Acute Mesenteric Ischemia (AMI) AMI is a rare and difficult-to-diagnose condition with high diagnostic delays and mortality rates. Its initial presentation often mimics sepsis or septic shock, leading to the early administration of broad-spectrum empirical antibiotics due to fears of bacterial translocation or perforation. Although surgical guidelines encourage systemic antibiotic use, there is insufficient evidence for its routine application.

Study Objective While data on the SeptiCyte LAB test is available for cardiac and digestive surgeries, there is none for vascular surgery. This study aims to evaluate the SeptiCyte LAB test's ability to identify postoperative SIRS patients to reduce empirical antibiotic use while awaiting standard bacteriology results and to assess the impact of surgery on the SeptiCyte LAB test. We will study patients admitted to intensive care units pre- and post-open laparotomy for the treatment of embolic or thrombotic AMI.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* Affiliated to health assurance system
* Hospitalized in the ICU for confirmed mesenteric ischemia* for less than 24 hours with an indication for laparotomy
* Hospitalized in the ICU for confirmed mesenteric ischemia* who underwent laparotomy for revascularization or digestive resection less than 24 hours ago
* Intraoperative bacteriological samples and blood cultures performed within 24 hours of medical management

Exclusion Criteria:

* decline to participate
* no consent available

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with suspected of confirmed acute mesenteric ischemia who required urgent surgery for revascularisation and/or intra-abdominal infection
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of bacterial coinfection during acute mesenteric ischemia | Day 0 (pre operative)
  Septicyte Lab test < 4 if there is no infection

SECONDARY OUTCOMES:
Diagnostic performance of Septicyte Lab test to rule out the presence of intra-abdominal infection during acute mesenteric ischemia | Day 0 (pre operative)
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value of the Septicyte Lab test
Diagnostic performance of PCT to rule out the presence of intra-abdominal infection during acute mesenteric ischemia | Day 0 (pre operative)
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value of the PCT
Diagnostic performance of CRP to rule out the presence of intra-abdominal infection during acute mesenteric ischemia | Day 0 (pre operative)
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value of the CRP
Change in Septicyte Lab test during the post-operative period to address the influence of surgery on the response of patient's immune system | Day 1
  Value of Septicyte Lab test

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No